CLINICAL TRIAL: NCT03593382
Title: Physiological and Behavioural Aspects of Insufficient Energy Availability in Females Endurance Athletes - Impact on Metabolism, Recovery and Health
Brief Title: Energy Availability in Female Athletes
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Lund University (Other); Herlev Hospital (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Other Study IDs: B285
Record Dates: First submitted 2012-09-16; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Female Athlete Triad
Keywords: Female endurance athletes; Energy Availability; Nutrient Availability; Bone Mineral Density; Menstrual dysfunction; Female athlete triad; Energy metabolism; Recovery after exercise; Endothelial function; Eating disorders; Performance
MeSH Terms: conditions — Female Athlete Triad Syndrome; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood Serum Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Female endurance athletes: Female endurance athletes recruited from Swedish and Danish national teams and competitive sport clubs

SUMMARY:
The purpose of this project is to study the impact of energy availability (EA) on female endurance athletes and the adaptive consequences of insufficient EA with a special reference to the impact on energy metabolism, reproductive-, vascular- and bone health as well as exercise capacity, neuromuscular performance, ability to recover from intense exercise and the genetic interaction.

Specific aims:

* To investigate the effects of EA on energy metabolism
* To investigate the effects of EA on reproductive, vascular- and bone health, and endocrine functions
* To investigate the effects of EA on exercise capacity
* To investigate the effects of EA on neuromuscular performance
* To investigate the effects of EA on recovery after exercise
* To identify potential dietary factors influencing EA, exercise capacity and neuromuscular performance
* To identify potential exercise factors influencing EA, exercise capacity and neuromuscular performance
* To identify potential psychological, behavoural and motivational aspects associated with insufficient EA

The investigators hypothesize that female athletes with insufficient energy availability have attenuated energy metabolism, reduced BMD, impaired endothelial function and decreased ability to recover between exercise bouts compared to matched controls with sufficient energy and nutrient intake. The investigators also hypothesize that EA influences exercise capacity and neuromuscular performance.

DETAILED DESCRIPTION:
The study population was recruited through the Danish and Swedish sport federations in weight-bearing endurance sports, and in local competitive endurance sports clubs, through flyers, webpage announcements and mailings. Interested athletes received the study protocol and a self-administered questionnaire, assessing age, sport, training regime, and self-assessed menstrual function. Athletes returning the questionnaire and who were interested in further participation were contacted by the research group. Before inclusion, all subjects were informed orally, and in writing, of all study procedures and signed an informed consent form. Subjects included and defined as elite endurance athletes were athletes at national team levels or competitive endurance athletes from regional sports clubs, 18-38 years of age, training a minimum of five times per week. Exclusion criteria included clinically verified menstrual dysfunction other than oligomenorrhea/functional hypothalamic amenorrhea; pregnancy; chronic illness; smoking; use of forms of contraceptives other than oral, e.g., hormonal coil/patches; inability or being unwilling to stop hormonal contraceptives for at least 6 weeks prior to investigation; or injuries preventing the athlete from training ≥ 2 weeks.

Data collection was performed on two consecutive days followed by a 7-day registration period in the athletes' normal environment. The first day comprised of examinations involving bone health, blood pressure and reproductive function. The second day included examinations of energy metabolism, aerobic capacity, as well as assessment of eating disorders. The subjects were instructed not to exercise for more than 30 min at low or moderate intensity on the day before, and on the first day of examination, and to arrive at the clinic in a fasted (from midnight) and rested state.

PROTOCOL OVERVIEW:

DAY 1: Start at 7:45 A.M.

1. Pragnancy test
2. Blood sampling
3. DXA scan
4. Blood pressure
5. Meal
6. Gynecological examination

DAY 2: Start at 7 A.M.

1. RMR
2. Blood sampling
3. Work efficiency
4. Meal
5. EDE interview
6. Incremental exercise test
7. EDI-questionnaire

7 DAY DIETARY AND ACTIVITY RECORD

The timing of the examination and registration period was planned individually for each subject in order to choose a period reflecting their habitual food habits and exercise regimes. Dietary intake and training intensity were recorded by the subjects for seven consecutive days to assess current EA. Energy intake was calculated from a prospective weighed (Exido 246030 Kitchen Scale, Gothenburg, Sweden) food record, using a nutrient analysis program, Dankost 2000 (Dankost, Copenhagen, Denmark) for Danish food items, and Dietist XP (Kost och Näringsdata AB, Bromma, Sweden) for Swedish food items. Subjects were given in-depth verbal and written instructions and a demonstration of how food and beverages should be weighed and registered. Subjects were instructed to maintain their normal food habits and eating patterns. Before entering data in the nutrient analysis program the same dietician reviewed all completed diet records and asked for supplementary information if needed, and the mean daily energy intake from the 7-day record was used in the analysis. In order to identify subjects who provided nutritional data of poor validity, the Goldberg cutoff was calculated using the equation described by Black (2000). Heart rate monitors (Polar RS400®, Stockholm, Sweden) and training logs were used to assess exercise energy expenditure. Subjects were instructed to maintain and to follow their normal training regime. They were, furthermore, instructed to describe each session in as much detail as possible, regarding type, duration, and intensity of exercise and to wear the heart rate monitor at all training sessions (except swimming) and during cycling (training as well as transportation).

Eating behavior was assessed using the Eating Disorder Inventory (EDI-3), a questionnaire assessing behavior and attitudes related to DE behavior, as well as to overt ED. Subjects were categorized as having DE behavior when the EDI risk subscale score for Drive for Thinness (DT) was ≥ 14, and/or a Body Dissatisfaction (BD) risk score ≥ 19 and without the presence of DSM-IV diagnosed ED. The Eating Disorder Examination (EDE-16) was used to determine whether subjects met the criteria for ED, according DSM-IVcriteria for anorexia nervosa, bulimia nervosa, and ED not otherwise specified (EDNOS). All interviews were performed by the same EDE-certified member of the research team.

Subjects were transported by car to the clinic on the morning of the second test day in order to minimize physical activity prior to the measurement. RMR was assessed between 7:00 and 8:30 h, after an overnight fast, using a ventilated open hood system (Oxycon Pro 4, Jeager, Germany). The system was automatically calibrated before each test, and again weekly, by an alcohol burning test with coefficients of variability (CV) of 0.7% for O2, 1.1% for CO2, 0.8%for the respiratory exchange ratio, and 2% for EE. After voiding, subjects laid down for 15 min before measurements of oxygen consumption (VO2) and carbon dioxide production (VCO2) over 35 min (the equation is defined under Calculations). Work efficiency was assessed by a standardized test protocol in the fasted state, initiated by the subject seated on the bicycle ergometer (Monark 939E, Monark Exercise AB, Vansbro, Sweden) for 6 min, followed by cycling for 6 min at 0W, 50W and 100W, respectively. An air-tight mask covering the mouth and nose was used in order to measure respiratory gas exchange (the equations for calculations are defined under Calculations). In order to calculate daily total EE, HR monitors (Polar RS400®) were used to assess EE during bicycle transportation, while actigraphy (ActiGraph GT3X®, Pensacola, FL, USA) and the data analysis software ActiLife 5 (ActiGraph) were used for assessment of NEAT. Subjects were instructed to wear an accelerometer on the wrist during sleep, and on the hip from getting up in the morning until bedtime, and only to take it off during showering, swimming, bicycle transportation, and training.

Two hours after a standardized breakfast, an incremental exercise test on the bicycle ergometer was performed, initiated by cycling for 6 min at 50W, followed by an increase in workload of 12-14 W/min until exhaustion. An air-tight mask covering the mouth and nose was used in order to measure VO2peak and respiratory exchange ratio, and HR (Polar RS400®) was measured.

Subjects using hormonal contraceptives were requested to stop for a minimum of 6 weeks prior to examination in order to secure a sufficientwashout period for exogenous estrogen and progesterone. Subjects not recovering their menstrual bleeding within the 6 weeks were contacted monthly by the research team during a follow-up period of a minimum of 3 months before gynecological assessment. Menstruating athletes were examined in the early follicular phase, on the third to fifth day of menstruation. A pregnancy test was performed on arrival at the hospital, and menstrual function was examined by an experienced gynecologist who performed a transvaginal ultrasound examination (Ultrasound Scanner, Class 1 type B, B-K Medical REF TYPE 2202, Bedfordshire, UK). The maximum number of ovarian follicles present in a single plane was counted, and total volume was assessed. Sex hormone status [estrogen, progesterone, LH, follicle stimulating hormone (FSH), sexual hormone binding globulin (SHBG), prolactin, dehydroepiandrosteron sulfate (DHEA-S), androstendion, and total testosterone] and anamnestic assessment, e.g., age of menarche, previous menstrual irregularities, use of hormonal contraceptives, and number of menstrual cycles during the last year, were recorded using the low EAin females questionnaire (LEAF-Q) (Melin et al., 2014). Subjects were then classified with eumenorrhea (menstrual cycles of 28 days ± 7 days and sex hormones within the normal range); oligomenorrhea (menstrual cycles > 35 days where other causes than hypothalamic suppression had been ruled out); FHA (either primary: no menarche after 15 years of age, or secondary: absence of at least three consecutive menstrual cycles where other causes than hypothalamic suppression had been ruled out) (Nattiv et al., 2007); other MDs (anatomic defects, hyperprolactinemia or other dysfunctional ovarian conditions); PCOS involving at least two of the following: (a) enlarged ovaries with a volume greater than 10 mL and/or ≥ one ovary demonstrating ≥ 12 follicles in one plane; (b) irregular or absence of bleeding; and (c) elevated androgen level, or otherwise androgen stigmatized.

Body weight was measured with an accuracy of 0.01 kg in underwear on an electronic scale (Lindeltronic 8000, Samhall Lavi AB, Kristianstad, Sweden). Height was measured without shoes and standing with legs together against a wall, using a fixed stadiometer (Hultafors AB, Hultafors, Sweden). After resting in a supine position for 7 min, HR and BP were measured three times (the mean was used) using an electronic sphygmomanometer (Microlife BP A100, Widnau, Switzerland). Hypotension was defined as a systolic BP < 90 mmHg and/or diastolic BP < 60 mmHg. Dual-energy X-ray absorptiometry (DXA) (Hologic, Model Discovery 2009, Hologic Inc.,Waltham, MA, USA) was used to determine fat-free, fat, and bone mass, respectively. BMD was determined for whole body, lumbar spine (L1-L4) and hip. All measurements and scans were performed in the fasted and resting state between 7:30 and 9:00 h, and were assessed by the same technician, and performed on the same scanner. Calibration of the Hologic Discovery 2009 was performed weekly, using a phantom provided by the manufacturer. Subjects were classified as having normal BMD: Z-scores > -1 in all measured sites, low BMD: Z-score -1 to -2 in at least one site, and osteoporosis: Z-score < -2 in at least one site together with minimum one secondary risk factor such as low EA, ED and oligomenorrhea/FHA.

Blood samples were drawn following an overnight fast from an antecubital vein on the first as well as on the second day, between 8:30 and 8:50 h, in a rested state.

ELIGIBILITY:
Inclusion Criteria:

* Female endurance athlete exercising at least 5 times/week

Exclusion Criteria:

* Exclusion criteria are:

  * Pregnancy
  * Metabolic disorders
  * Smoking
  * Use of psychopharmaca
  * Use of other forms of contraceptives than oral, e.g. hormonal coil or patches
  * Serious injury stopping the athlete from training ≥ 2 weeks.
  * Diabetes

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female endurance athletes exercising minimum 5 times a week will be recruited via the Danish and Swedish National Sport Federations (Team Danmark, Danmarks Idrætsforbund and Riksidrottsförbundet) and from competivite sport clubs.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Energy availability | Measurements performed once in the week after the two days of gynbaecological and physiological measurements
  Enenergy availability (kcal/kg FFM/day) was calculated as energy intake minus exercise energy expenditure relative to fat free mass based on the 7 day records of energy intake (kcal/day) and assessment of exercise energy expenditure (kcal/day) as well as the assessment of body composition at the first day of visit.

SECONDARY OUTCOMES:
Resting energy metabolism | Assessed once at the second visit which was between 6 weeks and 6 months after inclusion
  Resting metabolic rate (kcal/day and kcal/kg FFM/day by ventilated hood). RMR was assessed between 7:00 and 8:30 h, after an overnight fast, using a ventilated open hood system (Oxycon Pro 4, Jeager, Germany). The system was automatically calibrated before each test, and again weekly, by an alcohol burning test with coefficients of variability (CV) of 0.7% for O2, 1.1% for CO2, 0.8
  %for the respiratory exchange ratio, and 2% for EE. After voiding, subjects laid down for 15 min before measurements of oxygen consumption (VO2) and carbon dioxide production (VCO2) over 35 min.
Work efficiancy | Assessed once at the second visit which was between 6 weeks and 6 months after inclusion
  Work efficiency (energy metabolism during low intense exercise) (kcal/watt) efficiency was assessed by a standardized test protocol in the fasted state, initiated by the subject seated on the bicycle ergometer (Monark 939E, Monark Exercise AB, Vansbro, Sweden) for 6 min, followed by cycling for 6 min at 0W, 50W and 100W, respectively. An air-tight mask covering the mouth and nose was used in order to measure respiratory gas exchange.
Substrate utilisation | Substrate utilisation was assessed once at the second visit which was between 6 weeks and 6 months after inclusion
  Substrate utilization during and after exercise (O2 consumption and CO2 production, RQ)
Bone mineral content | Bone mineral content was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  Bone mineral content (g) was assessed via Dual-energy X-ray absorptiometry (DXA) (Hologic, Model Discovery 2009, Hologic Inc.,Waltham, MA, USA)
Bone mineral density | Bone mineral density was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  Bone mineral density (g/cm2) was assessed via Dual-energy X-ray absorptiometry (DXA) (Hologic, Model Discovery 2009, Hologic Inc.,Waltham, MA, USA)
Leptin | Leptin was assessed once at the first visit which was between 6 weeks and 6 months after inclusion.
  Leptin (ng/ml) Leptin was analyzed using Quantikine® ELISA (R&D Systems® Europe Ltd., Abingdon, UK). The lower analytic limit for leptin was 1.56 ng/mL; lower concentrations are associated with some uncertainty and therefore not automatically calculated. Blood samples were drawn following an overnight fast from an antecubital vein between 8:30 and 8:50 h, in a rested state.
Orthostatic blood pressure | Orthostatic blood pressure was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  Orthostatic blood pressure (mHg) reaction after moving from supine to standing position (tilt table from 0 to 70 degree)
Total cholesterols | Total cholesterol was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  Total cholesterols (mmol/L) was analyzed using VITROS Chemistry Products DT slides (Ortho-Clinical Diagnostics, Buckinghamshire, UK). Blood samples were drawn following an overnight fast from an antecubital vein between 8:30 and 8:50 h, in a rested state.
HDL cholesterol | HDL cholesterol was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  HDL (mmol/L) was analyzed using VITROS Chemistry Products DT slides (Ortho-Clinical Diagnostics, Buckinghamshire, UK). Blood samples were drawn following an overnight fast from an antecubital vein between 8:30 and 8:50 h, in a rested state.
LDL cholesterol | LDL cholesterol was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  LDL (mmol/L) was analyzed using VITROS Chemistry Products DT slides (Ortho-Clinical Diagnostics, Buckinghamshire, UK). Blood samples were drawn following an overnight fast from an antecubital vein between 8:30 and 8:50 h, in a rested state.
Eating Disorder Inventory-3 (EDI-3) | The subjects filled out the questionnaire once at the second visit which was between 6 weeks and 6 months after inclusion
  EDI-3 is a questionnaire assessing behavior and attitudes related to DE behavior, as well as to overt ED (12). Subjects were categorized as having DE behavior when the EDI risk subscale score for Drive for Thinness (DT) was ≥ 14, and/or a Body Dissatisfaction (BD) risk score ≥ 19, according the classification by Garner (2004) and without the presence of DSM-IV diagnosed ED.
Eating disorder examination-16 (EDE-16) clinical interview score | The interview was performed once at the second visit which was between 6 weeks and 6 months after inclusion
  The Eating Disorder Examination (EDE-16) is a validated semi-structured interview. It was used to determine whether subjects met the criteria for eating disorder, according to the DSM-IV criteria for anorexia nervosa, bulimia nervosa, and eating disorder not otherwise specified (EDNOS). All interviews were performed by the same EDE-certified member of the research team.
Low Energy Availability in Females Questionnaire (LEAF-Q) score | Subjects filled out the LEAF-Q once at the second visit which was between 6 weeks and 6 months after inclusion
  The LEAF-Q is a validated screening instrument for detecting low energy availability, assessing menstrual history, injuries and gastrointestinal function
Energy intake | Assessment of energy intake was performed once in the week after the two days of clinical examination
  Energy intake was assessed in order to calculate energy availability. Energy intake was calculated from a prospective weighed (Exido 246030 Kitchen Scale, Gothenburg, Sweden) food record, using a nutrient analysis program, Dankost 2000 (Dankost, Copenhagen, Denmark) for Danish food items, and Dietist XP (Kost och Näringsdata AB, Bromma, Sweden) for Swedish food items.
Exercise energy expenditure | Assessment of exercise energy expenditure was performed once in the week after the two days of examination
  Exercise energy expenditure was assessed in order to calculate energy availability. Heart rate monitors (Polar RS400®, Stockholm, Sweden) and training logs were used to assess exercise energy expenditure (EEE). Subjects were instructed to maintain and to follow their normal training regime. They were, furthermore, instructed to describe each session in as much detail as possible, regarding type, duration, and intensity of exercise and to wear the HR monitor at all training sessions (except swimming) and during cycling (training as well as transportation). The mean daily EEE for the sessions described as exercise by the subjects, was used and the method for calculation of current EA
Estrogen (estradiol) | Estradiol was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  Estradiol (pmol/L) was measured in order to assess reproductive function. Blood samples were drawn following an overnight fast from an antecubital vein between 8:30 and 8:50 h, in a rested state.
Follicle stimulating hormone (FSH) | FSH was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  FSH (IU/L) was measured in order to assess reproductive function. Blood samples were drawn following an overnight fast from an antecubital vein between 8:30 and 8:50 h, in a rested state.
Luteinizing hormone (LH) | LH was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  SHBG (nmol/L) was measured in order to assess reproductive function. Blood samples were drawn following an overnight fast from an antecubital vein between 8:30 and 8:50 h, in a rested state.
Prolactine | Prolactine was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  Prolactine (uIU/ml) was measured in order to assess reproductive function. Blood samples were drawn following an overnight fast from an antecubital vein between 8:30 and 8:50 h, in a rested state.
Sex hormone-binding globulin (SHBG) | SHBG was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  SHBG (nmol/L)
Total testosterone | Testosterone was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  Testosterone (nmol/L) was measured in order to assess reproductive function. Blood samples were drawn following an overnight fast from an antecubital vein between 8:30 and 8:50 h, in a rested state.
Dehydroepiandrosterone (DHEA) | DHEA was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  DHEA (µmol/L) was measured in order to assess reproductive function. Blood samples were drawn following an overnight fast from an antecubital vein between 8:30 and 8:50 h, in a rested state.
Training frequency | The training logs were applied by the subjects for 7 days following the two examination days
  Training frequency was assessed using a training log filled out by each participant
Training hours | The training logs wereapplied by the subjects for 7 days following the two examination days
  Training hours were assessed using a training log filled out by each participant
Reaction Time (RT) | RT was assessed 3 times at the second visit which was between 6 weeks and 6 months after inclusion
  After 10 min of rest, the reaction time (RT [ms]) test was performed on a portable computer connected to a linear encoder (MuscleLab 4010; Ergotest Innovation, Langensund, Norway). RT was assessed by measurement of time taken to press the space bar on the keyboard when the screen changed color while the finger rested on the space bar. After three trials for familiarization, the test procedure began. Each participant performed five reaction trials. The shortest RT of the five trials was used in the statistical analysis.
Knee Muscular Strentgh (KMS) | KMS was assessed 3 times at the second visit which was between 6 weeks and 6 months after inclusion
  Directly after the RT test, knee muscular strength (KMS [Nm]) measurements were performed using isokinetic dynamometry, and each participant performed strength tests using the right leg in a consistent order.
Knee Muscular Endurance (KME) | KME was assessed 3 times at the second visit which was between 6 weeks and 6 months after inclusion
  Directly after the RT test, knee muscular endurance (KME [w]) measurements were performed using isokinetic dynamometry, and each participant performed endurance tests using the right leg in a consistent order.
Non Exercise Activity Thermogenesis (NEAT) | The subjects wore the accelerometers for 7 days following the two examination days
  To assess NEAT (kcal/day) the data analysis software ActiLife 5 (ActiGraph) was used. Subjects were instructed to wear an accelerometer on the wrist during sleep, and on the hip from getting up in the morning until bedtime, and only to take it off during showering, swimming, bicycle transportation, and training.
Triglyceride | Triglyceride was assessed once at the first visit which was between 6 weeks and 6 months after inclusion
  Triglyceride (mmol/L) was analyzed using VITROS Chemistry Products DT slides (Ortho-Clinical Diagnostics, Buckinghamshire, UK).
Protein intake | Assessment of protein intake was performed once in the week after the two days of clinical examination
  Protein intake (g/day) was assessed from a prospective weighed (Exido 246030 Kitchen Scale, Gothenburg, Sweden) food record, using a nutrient analysis program, Dankost 2000 (Dankost, Copenhagen, Denmark) for Danish food items, and Dietist XP (Kost och Näringsdata AB, Bromma, Sweden) for Swedish food items.
Carbohydrate intake | Assessment of carbohydrate intake was performed once in the week after the two days of clinical examination
  Carbohydrate intake (g/day) was assessed from a prospective weighed (Exido 246030 Kitchen Scale, Gothenburg, Sweden) food record, using a nutrient analysis program, Dankost 2000 (Dankost, Copenhagen, Denmark) for Danish food items, and Dietist XP (Kost och Näringsdata AB, Bromma, Sweden) for Swedish food items.
Fat intake | Assessment of fat intake was performed once in the week after the two days of clinical examination
  Fat intake (g/day) was assessed from a prospective weighed (Exido 246030 Kitchen Scale, Gothenburg, Sweden) food record, using a nutrient analysis program, Dankost 2000 (Dankost, Copenhagen, Denmark) for Danish food items, and Dietist XP (Kost och Näringsdata AB, Bromma, Sweden) for Swedish food items.
Fiber intake | Assessment of fiber intake was performed once in the week after the two days of clinical examination
  Fiber intake (g/day) was assessed from a prospective weighed (Exido 246030 Kitchen Scale, Gothenburg, Sweden) food record, using a nutrient analysis program, Dankost 2000 (Dankost, Copenhagen, Denmark) for Danish food items, and Dietist XP (Kost och Näringsdata AB, Bromma, Sweden) for Swedish food items.

CONTACTS AND LOCATIONS:
Overall Officials: Anders sjödin, Assoc prof, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (3):
- Denmark (2):
  - Fertility Clinic Herlev Hospital, Herlev, Copenhagen
  - Department of Human Nutrition, Copenhagen
- Lund University, Lund, Skåne County, Sweden